CLINICAL TRIAL: NCT01921166
Title: Maximal Stimulation and Delayed Fertilization for Diminished Ovarian Reserve: a Randomized Pilot Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Diminished Ovarian Reserve
Record Dates: First submitted 2013-07-25; First posted 2013-08-13 (Estimated); Results first posted 2018-02-23 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2021-06

CONDITIONS: Infertility
Keywords: infertility; diminished ovarian reserve; fertilization in vitro; ovulation inducion; vitrification
MeSH Terms: conditions — Infertility | interventions — Clomiphene; Gonadotropins; Leuprolide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- clomiphene plus gonadotropins (Active Comparator): clomiphene plus gonadotropins
  Interventions: Drug: clomiphene plus gonadotropins
- Leuprolide flare (Active Comparator): Leuprolide flare
  Interventions: Drug: Leuprolide flare

INTERVENTIONS:
Drug: clomiphene plus gonadotropins — clomiphene plus gonadotropin ovulation induction
  Other Names: Clomid. Serophene. Gonal f. Bravelle. Follistim. Menopur.
  Arms: clomiphene plus gonadotropins
Drug: Leuprolide flare — Leuprolide flare ovulation induction
  Other Names: Lupron.
  Arms: Leuprolide flare

SUMMARY:
The purpose of the study is (A) to determine if the following novel approach improves the live birth rate with In-Vitro Fertilization (IVF) for women with a poor prognosis due to diminished ovarian reserve:

* ovarian stimulation with medications that are effective in women with diminished ovarian reserve but adversely affect the endometrium
* oocyte retrieval and vitrification
* fertilization and embryo transfer in a subsequent cycle with controlled endometrial preparation B) To determine the optimal stimulation protocol for women with diminished ovarian reserve incorporating oocyte vitrification

Women who are not eligible to participate in the Carolinas Medical Center (CMC) Assisted Reproductive Therapy program because of an extremely poor prognosis will be recruited for a prospective, randomized, open-label study to determine if a novel approach improves the live birth rate with traditional IVF "poor prognosis" stimulation protocols. The novel approach will incorporate one of two protocols utilizing medications that provide maximal ovarian stimulation but have a temporary detrimental fertility-reducing effect on the endometrium. If ovarian stimulation is adequate, oocyte retrieval will be performed and viable oocytes vitrified (stored in a "glass-like" state in liquid nitrogen). At a later time, oocyte warming and fertilization will be performed in a subsequent cycle, in which the endometrium has been prepared.

Key points include:

* Randomization to one of two ovarian stimulation protocols that have been shown to have a detrimental effect on the endometrium, and therefore are rarely used in a "fresh" IVF cycle
* Oocyte vitrification is considered to be an investigational procedure by the American Society of Reproductive Medicine (ASRM), and should only be performed under the supervision of an IRB. With oocyte vitrification, ovarian stimulation and oocyte retrieval can "unlinked" from embryo transfer, allowing embryo transfer to occur in a more optimal environment
* Endometrial preparation is routine for frozen embryo transfer

DETAILED DESCRIPTION:
Women who are not eligible to participate in the CMC Assisted Reproductive Therapy (ART) program because of an extremely poor prognosis will be recruited for a prospective, randomized, open-label study to determine if a novel approach improves the live birth rate with traditional IVF "poor prognosis" stimulation protocols. The novel approach will incorporate one of two protocols utilizing medications that provide maximal ovarian stimulation but have a temporary detrimental fertility-reducing effect on the endometrium. If ovarian stimulation is adequate, oocyte retrieval will be performed and viable oocytes vitrified (stored in a "glass-like" state in liquid nitrogen). At a later time, oocyte warming and fertilization will be performed in a subsequent cycle, in which the endometrium has been prepared.

Key points include:

* Randomization to one of two ovarian stimulation protocols that have been shown to have a detrimental effect on the endometrium, and therefore are rarely used in a "fresh" IVF cycle
* Oocyte vitrification is considered to be an investigational procedure by the American Society of Reproductive Medicine (ASRM), and should only be performed under the supervision of an IRB. With oocyte vitrification, ovarian stimulation and oocyte retrieval can be "unlinked" from embryo transfer, allowing embryo transfer to occur in a more optimal environment
* Endometrial preparation is routine for frozen embryo transfer Eligible patients will be randomized to one of two protocols: clomiphene + HMG or leuprolide flare protocol.

All subjects must undergo pre-cycle IVF testing as per routine for the CMC ART program. In general, the study will be comprised of subjects not eligible for IVF due to extremely poor prognosis because of expected compromised ovarian stimulation (see inclusion criteria below). Subjects are financially responsible for all treatments in this study. Randomized will be performed by a random number generator after informed consent has been signed. Randomization at this point will allow time to order and obtain required medications.

Cycle start requirements (performed cycle day 2 or 3):

* Basal Follicle Stimulating Hormone (FSH) 12 mIU/mL or less AND
* Basal estradiol 50 pg/mL or less AND
* Acceptable baseline ultrasound (no evidence of a condition for which IVF would be contraindicated) If patient does not meet start requirements, delay and repeat cycle start tests in the next IVF session.

Group 1: clomiphene + human menopausal gonadotropin Menopur ® (HMG)

* Clomiphene 100 mg cycle days 3-7 plus
* HMG 300 units daily beginning cycle day 3 and continued until day of HCG (Ovidrel) administration

Group 2: leuprolide flare + HMG

* leuprolide acetate 0.5 mg twice daily beginning cycle day 3 and continued until day of HCG (Ovidrel) administration
* HMG 300 units daily beginning cycle day 3 and continued until day of HCG (Ovidrel) administration

Both groups:

* Follow-up ultrasound, estradiol cycle day 8. Cancel cycle if estradiol is < 200 pg/mL. If estradiol is 200 pg/mL or higher, make HMG dose adjustments and schedule follow-up estradiol and ultrasound visits as per routine IVF protocol.
* Administer Ovidrel 500 mg when 2nd largest follicle reaches a mean diameter of 18mm. Cancel cycle if < 3 follicles 10mm or larger are recruited or if spontaneous ovulation occurs.
* Retrieval: per standard IVF routine
* Vitrification: all viable oocytes will be vitrified on the day of oocyte retrieval.
* Remainder of stimulation cycle: no additional medications
* Stimulation and retrieval cycle may be repeated at patient request if < 5 oocytes are vitrified to store additional oocytes for transfer cycle.

Transfer cycle:

* Programmed frozen embryo transfer protocol as per ART program routine: precycle treatment with oral contraceptives (OCP), leuprolide administration during OCP, OCP withdrawal bleeding, estrogen priming of endometrium, ultrasound assessment of endometrium after 12-14 days, addition of daily progesterone when endometrial thickness is 7mm or greater, oocyte warming/fertilization/transfer scheduled.
* Oocyte warming and intracytoplasmic sperm injection (ICSI): oocytes warmed on the 2nd day of progesterone administration (example, if progesterone is started on Monday, oocytes are warmed on Tuesday). Semen sample collected on day of warming and prepared per IVF routine for ICSI. Mature viable oocytes undergo ICSI. Per ART laboratory routine, oocytes are assessed for fertilization the following day. If embryos are available for transfer, the embryo transfer procedure is performed according to standard CMC ART program guidelines the 6-8 cell or blastocyst stage. If available, excess embryos may be cryopreserved, at patients' request, as per CMC ART Program routine. Follow-up hormonal therapy, pregnancy test(s), and ultrasound studies will be performed per CMC ART program protocol.

Vitrified oocytes will be discarded or kept in storage according to the terms of our oocyte storage agreement.

Crossover:

If a patient fails to conceive after the above, she may elect to cross-over into the opposite treatment group

ELIGIBILITY:
Inclusion Criteria:

* Basal FSH 17 IU/mL (highest ever)
* Basal FSH 15-17 (highest ever) and failed EFORT test
* Age > 43 at the time of expected retrieval
* Failure to conceive with a prior "poor prognosis" IVF stimulation protocol (microdose leuprolide flare or GnRH antagonist cycle) if administered because of evidence of diminished ovarian reserve
* Failure to conceive with 3 or more IVF cycles at CMC

Exclusion Criteria:

* Contraindications to IVF
* Contraindication to pregnancy
* Allergy or contraindication to medications used for IVF or embryo transfer
* Use for a gestational carrier
* Uncorrected or untreatable uterine infertility
* Smoking or substance abuse within 3 months of initiating stimulation for IVF

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2011-01; Primary Completion 2011-11 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bradley S Hurst, M.D., Principal Investigator — Wake Forest University Health Sciences

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Clomiphene Plus Gonadotropins | Leuprolide Flare
Started | 8 | 15
Completed | 8 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Clomiphene Plus Gonadotropins | Leuprolide Flare | Total
Number analyzed (Participants) | 8 | 15 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 15 | 23
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 15 | 23
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Oocytes
Description: Number of oocytes retrieved
Time Frame: up to 24 months
Measure: Number; unit: oocytes
Units Other Than Participants: oocytes
Arm/Group | Clomiphene Plus Gonadotropins | Leuprolide Flare
Number analyzed (Participants) | 8 | 15
Number analyzed (oocytes) | 19 | 47
oocytes | 19 | 47

2. Secondary Outcome: Number of Oocytes Vitrified
Time Frame: up to 24 months
Measure: Number; unit: oocytes
Arm/Group | Clomiphene Plus Gonadotropins | Leuprolide Flare
Number analyzed (Participants) | 8 | 15
oocytes | 19 | 47

3. Other Pre Specified Outcome: Number of Embryos From Vitrified Oocytes
Description: per ovarian stimulation treatment protocol
Time Frame: up to 24 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 24 months
Arm/Group | Clomiphene Plus Gonadotropins | Leuprolide Flare
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/15
Other Adverse Events (participants affected / at risk) | 0/8 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No